CLINICAL TRIAL: NCT05886595
Title: A 12-month Prospective Cohort Study of Mental Health Care Pathways of Adolescents and Young Adults
Brief Title: Being Young : My Mental Health
Acronym: JEMMA
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier St Anne (Other)
Collaborators: Groupement Interrégional de Recherche Clinique et d'Innovation (Other)
Responsible Party: Sponsor
Other Study IDs: D22-EPI031
Record Dates: First submitted 2023-05-09; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Mental Health Issue; Mental Disorder
Keywords: mental health; adolescent; young adult; psychiatry
MeSH Terms: conditions — Mental Disorders; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this prospective cohort study is to study the evolution of adolescent and young people's mental health over a 12-month period after presentation to an emergency department or crisis service for an acute psychiatric episode.

This study aims to:

* Describe the mental health care trajectories of adolescents and young adults after an acute psychiatric episode.
* Identify psychiatric disorders (such as anxiety, depression, eating disorders, suicidal thoughts, sleep, etc.) at the different time points of the study (at 3, 6, 9 and 12 months after inclusion) ;
* Assess the quality of life and functional capacity in daily activities of participants at each study time point ;
* Determine the socio-demographic, psychosocial and environmental factors associated with improving mental health over time and with mental health help seeking.

Patients aged from 10 to 24, presenting to one of the participating centers for an acute psychiatric episode, and who agree to participate, will be included in the study. Participants will have to complete an online questionnaire every 3 months over a 12-month period (at baseline (T0), at 3 months (T3), at 6 months (T6), at 9 month (T9) and at 12 months (T12))

DETAILED DESCRIPTION:
Recruitment process

A poster campaign will be carry out in all study locations. Patients aged between 10 and 25 visiting one of the study location will be invited to participate in the study. The clinical research associates will visit all study location on a weekly basis in order to present the study to eligible patients.

After checking the inclusion criteria, the clinical research associate will call eligible patients (or their legal representative for patients under 18) to present the study, the implications related to study participation, and obtain their oral consent. Patients who were willing to participate in the study will be automatically identify by a number.

Follow-up :

Patients will have to complete an online questionnaire at different time of the study: at baseline, at 3 months, at 6 months, at 9 months and at 12 months. For the participants aged under 18, the questionnaire will have to complete by or with the help of the parental representative.

Investigators will collect socio-demographic, clinical data related to the acute psychiatric episode, and health care pathway over time. Mental health assessments will be based on standardized questionnaires.

Clinical research associates will send an email to all participants to complete the initial questionnaire (at baseline). Then, they will coordinate patient follow-up, and will send automatic reminder through email at the different times of the study :at 3 months (M3), 6 months (M6), 9 months (M9) and 12 months (M12) to complete the follow-up questionnaires online. Patients will be awarded a gift voucher worth €10 after each completed questionnaire.

ELIGIBILITY:
Inclusion Criteria :

All patients

* aged from 10 to 24 years old
* had an consultation in one the study locations for psychiatric reason

Exclusion Criteria :

* Absence of consent of the patient or the parental authority holder (for minor patient)
* Adult patients under legal protection
* Lack of proficiency in French (language of the study)

Ages: 10 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population focuses on patient aged between 10 and 24 years old who have reached out to a mental health care service selected as a study location.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-09-04 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Strengths and Difficulties Questionnaire (SDQ) | Baseline
  brief emotional and behavioural screening questionnaire for children and young people Minimal value : From Not True Maximum value : Certainly True
Strengths and Difficulties Questionnaire (SDQ) | Month 3
  brief emotional and behavioural screening questionnaire for children and young people at month 3 Minimal value : From Not True Maximum value : Certainly True
Strengths and Difficulties Questionnaire (SDQ) | Month 6
  brief emotional and behavioural screening questionnaire for children and young people at month 6 Minimal value : From Not True Maximum value : Certainly True
Strengths and Difficulties Questionnaire (SDQ) | Month 9
  brief emotional and behavioural screening questionnaire for children and young people at month 9 Minimal value : From Not True Maximum value : Certainly True
Strengths and Difficulties Questionnaire (SDQ) | Month 12
  brief emotional and behavioural screening questionnaire for children and young people at month 12 Minimal value : From Not True Maximum value : Certainly True

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | baseline
  Measuring tool for anxiety and depression in a general medical population of patients at baseline 0-7 = Normal, 8-10 =Borderline abnormal (borderline case), 11-21 = Abnormal(case)
Hospital Anxiety and Depression Scale (HADS) | Month 3
  Measuring tool for anxiety and depression in a general medical population of patients at month 3 0-7 = Normal, 8-10 =Borderline abnormal (borderline case), 11-21 = Abnormal(case)
Hospital Anxiety and Depression Scale (HADS) | Month 6
  Measuring tool for anxiety and depression in a general medical population of patients at month 6 0-7 = Normal, 8-10 =Borderline abnormal (borderline case), 11-21 = Abnormal(case)
Hospital Anxiety and Depression Scale (HADS) | Month 9
  Measuring tool for anxiety and depression in a general medical population of patients at month 9 0-7 = Normal, 8-10 =Borderline abnormal (borderline case), 11-21 = Abnormal(case)
Hospital Anxiety and Depression Scale (HADS) | Month 12
  Measuring tool for anxiety and depression in a general medical population of patients at month 12 0-7 = Normal, 8-10 =Borderline abnormal (borderline case), 11-21 = Abnormal(case)
Suicidal Behaviors Questionnaire (SBQ) | baseline
  Self report questionnaire to identify risk factors for suicide in adolescents and adults.
  Scale from 0= I never had this thought to 6= Almost everyday
Suicidal Behaviors Questionnaire (SBQ) | month 3
  Self report questionnaire to identify risk factors for suicide in adolescents and adults at month 3 Scale from Scale from 0= I never had this thought to 6= Almost everyday
Suicidal Behaviors Questionnaire (SBQ) | month 6
  Self report questionnaire to identify risk factors for suicide in adolescents and adults at month 6 Scale from 0= I never had this thought to 6= Almost everyday
Suicidal Behaviors Questionnaire (SBQ) | month 9
  Self report questionnaire to identify risk factors for suicide in adolescents and adults at month 9 scale from 0= I never had this thought to 6= Almost everyday
Suicidal Behaviors Questionnaire (SBQ) | month 12
  Self report questionnaire to identify risk factors for suicide in adolescents and adults at month 12 scale from 0= I never had this thought to 6= Almost everyday
Ask Suicide-Screening Questions (ASQ) | baseline
  Screening tool to identify individuals that require further mental health/suicide safety assessment at baseline Yes or No scale If patient answers "No" to all questions 1 through 4, screening is complete (not necessary to ask question #5) If patient answers "Yes" to any of questions or refuses to answer, they are considered a positive screen.
Ask Suicide-Screening Questions (ASQ) | month 3
  Screening tool to identify individuals that require further mental health/suicide safety assessment at month 3 Yes or No scale If patient answers "No" to all questions 1 through 4, screening is complete (not necessary to ask question #5) If patient answers "Yes" to any of questions or refuses to answer, they are considered a positive screen.
Ask Suicide-Screening Questions (ASQ) | month 6
  Screening tool to identify individuals that require further mental health/suicide safety assessment at month 6 Yes or No scale If patient answers "No" to all questions 1 through 4, screening is complete (not necessary to ask question #5) If patient answers "Yes" to any of questions or refuses to answer, they are considered a positive screen.
Ask Suicide-Screening Questions (ASQ) | month 9
  Screening tool to identify individuals that require further mental health/suicide safety assessment at month 9 Yes or No scale If patient answers "No" to all questions 1 through 4, screening is complete (not necessary to ask question #5) If patient answers "Yes" to any of questions or refuses to answer, they are considered a positive screen.
Ask Suicide-Screening Questions (ASQ) | month 12
  Screening tool to identify individuals that require further mental health/suicide safety assessment at month 12 Yes or No scale If patient answers "No" to all questions 1 through 4, screening is complete (not necessary to ask question #5) If patient answers "Yes" to any of questions or refuses to answer, they are considered a positive screen.
Addictive disorders | baseline
  Questionnaire on alcohol and psychoactive substances consumption at baseline
Addictive disorders | month 3
  Questionnaire on alcohol and psychoactive substances consumption at month 3
Addictive disorders | month 6
  Questionnaire on alcohol and psychoactive substances consumption at month 6
Addictive disorders | month 9
  Questionnaire on alcohol and psychoactive substances consumption at month 9
Addictive disorders | month 12
  Questionnaire on alcohol and psychoactive substances consumption at month 12
Quality of Life, Enjoyment, and Satisfaction Questionnaire- (Q-LES-Q) | baseline
  self-report measure designed to obtain sensitive measures of the degree of enjoyment and satisfaction experienced in various areas of daily functioning in adults at baseline 5-point scale from 1 (Very Poor) to 5 (Very Good)
Quality of Life, Enjoyment, and Satisfaction Questionnaire- (Q-LES-Q) | month 3
  self-report measure designed to obtain sensitive measures of the degree of enjoyment and satisfaction experienced in various areas of daily functioning in adults at month 3 5-point scale from 1 (Very Poor) to 5 (Very Good)
Quality of Life, Enjoyment, and Satisfaction Questionnaire- (Q-LES-Q) | month 6
  self-report measure designed to obtain sensitive measures of the degree of enjoyment and satisfaction experienced in various areas of daily functioning in adults at month 6 5-point scale from 1 (Very Poor) to 5 (Very Good)
Quality of Life, Enjoyment, and Satisfaction Questionnaire- (Q-LES-Q) | month 9
  self-report measure designed to obtain sensitive measures of the degree of enjoyment and satisfaction experienced in various areas of daily functioning in adults at month 9 5-point scale from 1 (Very Poor) to 5 (Very Good)
Quality of Life, Enjoyment, and Satisfaction Questionnaire- (Q-LES-Q) | month 12
  self-report measure designed to obtain sensitive measures of the degree of enjoyment and satisfaction experienced in various areas of daily functioning in adults at month 12 5-point scale from 1 (Very Poor) to 5 (Very Good)
Pediatric Quality of Life Enjoyment and Satisfaction Questionnaire (P-Q-LES-Q) | baseline
  self-report measure designed to obtain sensitive measures of the degree of enjoyment and satisfaction experienced in various areas of daily functioning in children at baseline 5-point scale from 1 (Very Poor) to 5 (Very Good)
Pediatric Quality of Life Enjoyment and Satisfaction Questionnaire (P-Q-LES-Q) | month 3
  self-report measure designed to obtain sensitive measures of the degree of enjoyment and satisfaction experienced in various areas of daily functioning in children at month 3 5-point scale from 1 (Very Poor) to 5 (Very Good)
Pediatric Quality of Life Enjoyment and Satisfaction Questionnaire (P-Q-LES-Q) | month 6
  self-report measure designed to obtain sensitive measures of the degree of enjoyment and satisfaction experienced in various areas of daily functioning in children at month 6 5-point scale from 1 (Very Poor) to 5 (Very Good)
Pediatric Quality of Life Enjoyment and Satisfaction Questionnaire (P-Q-LES-Q) | month 9
  self-report measure designed to obtain sensitive measures of the degree of enjoyment and satisfaction experienced in various areas of daily functioning in children at month 9 5-point scale from 1 (Very Poor) to 5 (Very Good)
Pediatric Quality of Life Enjoyment and Satisfaction Questionnaire (P-Q-LES-Q) | month 12
  self-report measure designed to obtain sensitive measures of the degree of enjoyment and satisfaction experienced in various areas of daily functioning in children at month 12 5-point scale from 1 (Very Poor) to 5 (Very Good)
Sleep disorders | baseline
  Questionnaire on difficulties that affect children and adults' sleep patterns at baseline
Sleep disorders | month 3
  Questionnaire on difficulties affecting children and adults' sleep patterns at month 3
Sleep disorders | month 6
  Questionnaire on difficulties affecting children and adults' sleep patterns at month 6
Sleep disorders | month 9
  Questionnaire on difficulties affecting children and adults' sleep patterns at month 9
Sleep disorders | month 12
  questionnaire on difficulties affecting children and adults' sleep patterns at month 12
Patient healthcare trajectory | baseline
  Questionnaire on the type of health care professional, the mental health care services visited,the frequency of medical appointments, the health events (hospitalization, emergency unit, suicide attempt) at baseline
Patient healthcare trajectory | month 3
  Questionnaire on the type of health care professional, the mental health care services visited,the frequency of medical appointments, the health events (hospitalization, emergency unit, suicide attempt) at month 3
Patient healthcare trajectory | month 6
  Questionnaire on the type of health care professional, the mental health care services visited,the frequency of medical appointments, the health events (hospitalization, emergency unit, suicide attempt) at month 6
Patient healthcare trajectory | month 9
  Questionnaire on the type of health care professional, the mental health care services visited,the frequency of medical appointments, the health events (hospitalization, emergency unit, suicide attempt) at month 9
Patient healthcare trajectory | month 12
  Questionnaire on the type of health care professional, the mental health care services visited,the frequency of medical appointments, the health events (hospitalization, emergency unit, suicide attempt) at month 12
social relation, social integration and social support | baseline
  questionnaire on difficulties related to social relation, social integration and social support affecting children and adult' mental health at baseline
social relation, social integration and social support | month 3
  questionnaire on difficulties related to social relation, social integration and social support affecting children and adult' mental health at month 3
social relation, social integration and social support | month 6
  questionnaire on difficulties related to social relation, social integration and social support affecting children and adult' mental health at month 6
social relation, social integration and social support | month 9
  questionnaire on difficulties related to social relation, social integration and social support affecting children and adult' mental health at month 9
social relation, social integration and social support | month 12
  questionnaire on difficulties related to social relation, social integration and social support affecting children and adult' mental health at month 12
sociodemographic , environmental and psycho social factors | baseline
  socio-demographic variables questionnaire (age, sex, education, household, employment or schooling, income, health insurance, medical history, psychiatric history if any) at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle SABBAH-LIM, Pediatric psychiatrist, Principal Investigator — GHU Paris Psychiatrie et Neurosciences
Locations (7):
- France (7):
  - Pediatric Emergency Department - Armand Trousseau Hospital, Paris, Île-de-France Region
  - ATRAP (Acute unit for child outpatients), Paris, Île-de-France Region
  - C.P.O.A (Psychiatric Emergency Department), Paris, Île-de-France Region
  - Pediatric Emergency Department - Necker Hospital, Paris, Île-de-France Region
  - CIAPA (Inpatient unit for Adolescents), Paris, Île-de-France Region
  - Adult Emergency Department - Bichât Hospital, Paris, Île-de-France Region
  - Pediatric Emergency Department - Robert Debré Hospital, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Undecided